CLINICAL TRIAL: NCT00791518
Title: An Evaluation of Lung Function and Symptoms in Patients With Chronic Obstructive Pulmonary Disease (COPD) on Long-Acting Bronchodilator Monotherapy
Brief Title: Evaluation of Lung Function and Symptoms in Patients Diagnosed With Chronic Obstructive Pulmonary Disease (COPD) on Long-Acting Bronchodilator Monotherapy
Acronym: LABD
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111891
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2010-04-22 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No group: No group
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — No intervention

SUMMARY:
A multicenter study to evaluate lung function and symptoms in subjects with COPD who have been on regular use of only one long-acting bronchodilator.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smoking history-Current or ex-smokers (defined as stopped smoking for at least three months prior to the study visit)
* Established history of COPD as diagnosed by a physician
* Regular use (prescribed for use every day) of only one long-acting bronchodilator greater than or equal to one month before the study visit
* Ability to read, comprehend, and record information in the English language

Exclusion Criteria:

* Currently active asthma (receiving asthma therapy and or having asthma symptoms)
* Use of ipratropium/albuterol combination products greater than three times per day, use of inhaled corticosteroids, use of inhaled corticosteroid/long-acting beta-agonist combinations, theophylline preparations, or oral beta agonists within 3 months prior to the study visit
* Previous lung surgery
* Other respiratory disorders other than COPD
* Current alcohol, illegal drug, or solvent abuse
* Females with a positive urine pregnancy test at the study visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed COPD who are on only one long acting bronchodilator medication to control their COPD symptoms.
Sampling Method: Probability Sample
Enrollment: 1084 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- United States (54):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Naranja, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Biddeford, Maine
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Clairton, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Milan, Tennessee
  - GSK Investigational Site, New Tazewell, Tennessee
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Wichita Falls, Texas

REFERENCES:
- [Background] Dransfield MT, Bailey W, Crater G, Emmett A, O'Dell DM, Yawn B. Disease severity and symptoms among patients receiving monotherapy for COPD. Prim Care Respir J. 2011 Mar;20(1):46-53. doi: 10.4104/pcrj.2010.00059. PMID 20886200

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Diagnosed COPD: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician
Period: Overall Study
Arm/Group | Participants With Diagnosed COPD
Started | 1084
Completed | 991
Not Completed | 93
Not completed — Protocol Violation | 93

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Diagnosed COPD
Number analyzed (Participants) | 1084
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 537
  Male | 547
Race/Ethnicity, Customized [Number; unit: participants] — One participant chose more than one race category; this participant was counted twice.
  participants
    White | 933
    African American/African Heritage | 146
    American Indian or Alaska Native | 3
    Asian | 1
    Japanese East Asian Heritage | 1
    American Indian or Alaska Native and White | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Whose Post-albuterol Forced Expiratory Volume in One Second (FEV1) Was <80% Predicted Normal
Description: The percentage of participants on long-acting bronchodilator (LABD) monotherapy who had a post-albuterol FEV1) <80% predicted normal was calculated. FEV1 is the amount of air that can be expelled from the lungs in one second after a full inspiration. Predicted normal values for FEV1 were calculated using the reference values from the third National Health and Nutrition Examination Survey (NHANES III). Values are based on the participants' age, height, sex, and race; thus, normal values vary based on participants' demographics.
Time Frame: Day 1 of a 1-day study; 15-30 min post-albuterol (self-administered)
Population: All participants enrolled in the study who had a post-albuterol FEV1 measurement. Some participants had unacceptable post-albuterol spirometry measurements and were not included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Diagnosed COPD
Number analyzed (Participants) | 1072
percentage of participants
  <80% predicted normal | 70
  >=80% predicted normal | 30

2. Secondary Outcome: Percentage of Participants Whose Post-albuterol FEV1 Was <50% Predicted Normal
Description: The percentage of participants on long-acting bronchodilator (LABD) monotherapy who met spirometric criteria for chronic obstructive pulmonary disease (COPD) and who had a post-albuterol FEV1 (the amount of air expelled from the lungs in one second after a full inspiration) <50% predicted normal was calculated. Predicted normal values for FEV1 were calculated using the reference values from the third National Health and Nutrition Examination Survey (NHANES III). Values are based on the participants' age, height, sex, and race; thus, normal values vary based on participants' demographics.
Time Frame: Day 1 of a 1-day study; 15-30 min post-albuterol (self-administered)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Diagnosed COPD
Number analyzed (Participants) | 1072
percentage of participants
  <50% predicted normal | 23
  >=50% predicted normal | 77

3. Secondary Outcome: Number of Participants With the Categorized Post-albuterol Forced Expiratory Volume in One Second/Forced Vital Capacity (FEV1/FVC) Ratios
Description: The ratio is calculated as the amount of air expelled from the lungs in one second after a full inspiration (FEV1) divided by the volume of air that can forcibly be blown out after a full inspiration (FVC).
Time Frame: Day 1 of a 1-day study
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants With Diagnosed COPD
Number analyzed (Participants) | 1072
participants
  <=0.70 | 689
  >0.70 | 383

4. Secondary Outcome: Mean Modified Medical Research Council (mMRC) Dyspnea Scale Scores for Participants With Post-albuterol FEV1 <80% and >=80%
Description: The 5-point mMRC Dyspnea Scale measures the level of dyspnea (trouble breathing) experienced by participants. Scores range from 0 (none) to 4 (very severe).
Time Frame: Day 1 of a 1-day study
Population: All participants enrolled in the study who had an mMRC score with post-albuterol FEV1 <80% and >=80% percent predicted
Measure: Mean (Standard Error); unit: points on a scale
Groups:
- Participants With Diagnosed COPD and Post-albuterol FEV1 <80%: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician who also had a post-albuterol FEV1 <80%
- Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician who also had a post-albuterol FEV1 >=80%
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <80% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%
Number analyzed (Participants) | 754 | 318
points on a scale | 1.7 (0.04) | 1.6 (0.05)
Statistical Analysis 1: Comparison: Participants With Diagnosed COPD and Post-albuterol FEV1 <80% vs Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%; Test type: Superiority or Other; Least squares mean difference = 0.2, 95% CI [0.1 to 0.4] — Least squares mean differences are calculated as <80% group minus >=80% group and are adjusted for Investigator

5. Secondary Outcome: Mean mMRC Dyspnea Scale Scores for Participants With Post-albuterol FEV1 <50% and >=50%
Description: as for outcome 4
Time Frame: Day 1 of a 1-day study
Population: All participants enrolled in the study who had an mMRC score with post-albuterol FEV1 <50% and >=50% predicted
Measure: Mean (Standard Error); unit: points on a scale
Groups:
- Participants With Diagnosed COPD and Post-albuterol FEV1 <50%: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician who also had a post-albuterol FEV1 <50%
- Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician who also had a post-albuterol FEV1 >=80%
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <50% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%
Number analyzed (Participants) | 242 | 819
points on a scale | 1.9 (0.06) | 1.6 (0.03)
Statistical Analysis 1: Comparison: Participants With Diagnosed COPD and Post-albuterol FEV1 <50% vs Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%; Test type: Superiority or Other; Least squares mean difference = 0.3, 95% CI [0.2 to 0.4] — Least squares mean differences are calculated as <50% group minus >=50% group and was adjusted for Investigator

6. Secondary Outcome: Number of Participants Who Had a COPD Exacerbation Requiring Hospitalization With Post-albuterol FEV1 <80% and >=80%
Description: The number of participants who had a COPD exacerbation (defined as worsening of COPD symptoms) requiring hospitalization was calculated.
Time Frame: Day 1 of a 1-day study
Population: All participants enrolled in the study who had an acceptable post-albuterol FEV1 measure
Measure: Number; unit: participants
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <80% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%
Number analyzed (Participants) | 754 | 318
participants | 41 | 7

7. Secondary Outcome: Number of Participants Who Had a COPD Exacerbation Requiring Hospitalization With Post-albuterol FEV1 <50% and >=50%
Description: as for outcome 6
Time Frame: Day 1 of 1-day study
Population: All participants enrolled in the study who had an acceptable post-albuterol FEV1 measure
Measure: Number; unit: participants
Groups:
- Participants With Diagnosed COPD and Post-albuterol FEV1 <50%: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician and a post-albuterol FEV1 <50%
- Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician and a post-albuterol FEV1 >=50%
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <50% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%
Number analyzed (Participants) | 244 | 828
participants | 16 | 32

8. Secondary Outcome: Number of Participants Who Had a COPD Exacerbation Requiring Oral Corticosteroids and/or Antibiotics With Post-albuterol FEV1 <80% and >=80%
Description: The number of participants with a COPD exacerbation (worsening of COPD symptoms) requiring treatment with oral corticosteroids and/or antibiotics was calculated.
Time Frame: Day 1 of 1-day study
Population: All participants enrolled in the study who had an acceptable post-albuterol FEV1 measure
Measure: Number; unit: participants
Groups:
- Participants With Diagnosed COPD and Post-albuterol FEV1 <80%: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician with a post-albuterol FEV1 <80%
- Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%: Current and previous smokers with at least a 10 pack/year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician with a post-albuterol FEV1 >=80%
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <80% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%
Number analyzed (Participants) | 754 | 318
participants | 246 | 117

9. Secondary Outcome: Number of Participants Who Had a COPD Exacerbation Requiring Oral Corticosteroids and/or Antibiotics With Post-albuterol FEV1 <50% and >=50%
Description: as for outcome 8
Time Frame: Day 1 of 1-day study
Population: All participants enrolled in the study who had an acceptable post-albuterol FEV1 measure
Measure: Number; unit: participants
Groups:
- Participants With Diagnosed COPD and Post-albuterol FEV1 <50%: Current and previous smokers with at least a 10 pack/-year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician with a post-albuterol FEV1 <50%
- Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%: Current and previous smokers with at least a 10 pack/-year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician with a post-albuterol FEV1 >=50%
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <50% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%
Number analyzed (Participants) | 244 | 828
participants | 79 | 284

10. Secondary Outcome: Mean Puffs From All Short-acting Bronchodilators Used in the Past Two Weeks in Participants With an FEV1 of <80% and >=80%
Description: The average number of puffs from all short-acting bronchodilators used in the past 2 weeks was calculated.
Time Frame: Day 1 of a 1-day study
Population: All participants enrolled in the study who had an acceptable post-albuterol FEV1 measure
Measure: Mean (Standard Error); unit: puffs
Groups:
- Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%: Current and previous smokers with at least a 10 pack/-year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician with a post-albuterol FEV1 >=80%
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <80% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%
Number analyzed (Participants) | 754 | 318
puffs | 3.8 (0.33) | 2.3 (0.43)
Statistical Analysis 1: Comparison: Participants With Diagnosed COPD and Post-albuterol FEV1 <80% vs Participants With Diagnosed COPD and Post-albuterol FEV1 >=80%; Test type: Superiority or Other; Least squares mean difference = 0.7, 95% CI [-0.4 to 1.7] — Least squares mean differences are calculated as <80% group minus >=80% group and was adjusted for Investigator

11. Secondary Outcome: Mean Number of Puffs From All Short-acting Bronchodilators Used in the Past Two Weeks in Participants With an FEV1 of <50% and >=50%
Description: The average number of puffs from all short-acting bronchodilators used in the past 2 weeks was calculated.
Time Frame: Day 1 of a 1-day study
Population: All participants enrolled in the study who had an acceptable post-albuterol FEV1 measure
Measure: Mean (Standard Error); unit: puffs
Groups:
- Participants With Diagnosed COPD and Post-albuterol FEV1 <50%: Current and previous smokers with at least a 10 pack-year history of cigarette smoking and an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician with a post-albuterol FEV1 <50%
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <50% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%
Number analyzed (Participants) | 244 | 828
puffs | 5.2 (0.66) | 2.8 (0.28)
Statistical Analysis 1: Comparison: Participants With Diagnosed COPD and Post-albuterol FEV1 <50% vs Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%; Test type: Superiority or Other; Least squares mean difference = 0.9, 95% CI [-0.2 to 2.1] — Least squares mean differences are calculated as <50% group minus >=50% group and was adjusted for Investigator

12. Secondary Outcome: Number of Participants With Reports of Diagnosis and/or Treatment for Specific Cardiovascular (Heart), Psychiatric (Anxiety or Depression), and/or Bone Disorders in the <80%, >=80%, <50%, and >=50% FEV1 Groups
Description: The number of participants with the indicated affected medical conditions were counted.
Time Frame: Day 1 of a 1-day study
Population: All participants enrolled in the study who had an acceptable post-albuterol FEV1 measure
Measure: Number; unit: participants
Groups:
- Participants With Diagnosed COPD and Post-albuterol FEV1 <80%: Current and previous smokers with at least a 10 pack/-year history of cigarette smoking and a an established history of chronic obstructive pulmonary disease (COPD) as diagnosed by a physician with a post-albuterol FEV1 <80%
Arm/Group | Participants With Diagnosed COPD and Post-albuterol FEV1 <80% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=80% | Participants With Diagnosed COPD and Post-albuterol FEV1 <50% | Participants With Diagnosed COPD and Post-albuterol FEV1 >=50%
Number analyzed (Participants) | 754 | 318 | 244 | 828
participants
  Hypertension | 389 | 134 | 123 | 400
  Coronary artery disease | 87 | 24 | 26 | 85
  Edema | 69 | 9 | 23 | 55
  Atherosclerosis | 50 | 11 | 20 | 41
  Arrhythmia | 40 | 16 | 16 | 40
  Heart failure | 26 | 7 | 10 | 23
  Stable angina | 25 | 7 | 13 | 19
  Peripheral vascular disease | 22 | 9 | 6 | 25
  Valvular heart disease | 18 | 7 | 6 | 19
  Pulmonary edema | 11 | 4 | 6 | 9
  Ischemic heart disease without cardiomyopathy | 10 | 2 | 5 | 7
  Cardiomyopathy | 8 | 3 | 4 | 7
  Ischemic heart disease with cardiomyopathy | 11 | 0 | 5 | 6
  Cardiomegaly | 8 | 1 | 3 | 6
  Left ventricular dysfunction | 5 | 3 | 1 | 7
  Diastolic dysfunction | 5 | 2 | 1 | 6
  Cerebrovascular disease | 5 | 0 | 2 | 3
  Left ventricular hypertrophy | 4 | 1 | 2 | 3
  Stroke | 1 | 3 | 0 | 4
  Cardiac arrest | 2 | 1 | 0 | 3
  Myocardial infarction | 1 | 1 | 1 | 1
  Transient ischemic attack | 0 | 2 | 0 | 2
  Unstable angina | 2 | 0 | 0 | 2
  Generalized anxiety disorder | 113 | 38 | 37 | 114
  Major depressive disorder, recurrent episode | 107 | 45 | 30 | 122
  Social anxiety disorder (social phobia) | 24 | 17 | 7 | 34
  Panic disorder | 24 | 12 | 7 | 29
  Major depressive disorder, single episode | 17 | 6 | 4 | 19
  Post-traumatic stress disorder | 14 | 8 | 4 | 18
  Attention deficit/hyperactivity disorder | 9 | 4 | 4 | 9
  Osteoporosis | 92 | 26 | 29 | 89
  Osteopenia | 32 | 10 | 11 | 31

ADVERSE EVENTS:
Time Frame: Day 1 of a 1-day study
Arm/Group | Participants With Diagnosed COPD
Serious Adverse Events (participants affected / at risk) | 0/1084
Other Adverse Events (participants affected / at risk) | 5/1084
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Diagnosed COPD (N=1084)
Tooth fracture (Injury, poisoning and procedural complications) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Tremor (Nervous system disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.